CLINICAL TRIAL: NCT05844800
Title: The Effect of Surgical Repair of Chest on Postural Stability Among Patients With Pectus Excavatum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Wielkopolska Centre of Pulmonology and Thoracic Surgery in Poznan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Maria Jarosz PhD Thesis
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Pectus Excavatum
Keywords: Pectus Excavatum; Postural Stability
MeSH Terms: conditions — Funnel Chest | interventions — Anesthesia, Epidural; Bupivacaine

STUDY DESIGN:
Intervention Model Description: The experimental group of pectus excavatum patients (n=21) pre- and post intervention examination and control group of healthy subjects (n=22) examined twice.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectus Excavatum (Experimental): Patients included in the study after preoperative examination underwent the Nuss surgery procedure - a minimally-invasive repair technique of Pectus Excavatum (MIRPE)
  Interventions: Procedure: Nuss repair of Pectus Excavatum; Drug: Epidural anesthesia
- Healthy Control (No Intervention): Healthy control group with no posture defects

INTERVENTIONS:
Procedure: Nuss repair of Pectus Excavatum — The Nuss procedure is a minimally-invasive repair technique of PE (MIRPE), whereby one to three curved metal bars are inserted behind the sternum to correct the shape of the anterior chest wall. The bars are left in situ for three years and then removed.
  Other Names: minimally-invasive repair technique of Pectus Excavatum (MIRPE)
  Arms: Pectus Excavatum
Drug: Epidural anesthesia — The Nuss procedure of pectus excavatum repair surgery is performed under general anesthesia. Epidural anesthesia, with a constant infusion of 0.25% bupivacaine, was routinely used and was maintained in the early postoperative period.
  Other Names: Bupivacaine
  Arms: Pectus Excavatum

SUMMARY:
The goal of this study is to determine the effect of Nuss minimally-invasive repair technique of pectus excavatum (PE) on the postural stability in patients with PE.

The main questions it aims to answer are:

* How surgical chest wall repair will affect postural stability of PE patients?
* What is the difference in postural stability between patients with PE and healthy controls? Participants will undergo the Nuss repair surgery and will be tested before and afterwards for their postural stability with the use of the posturography method.

Researchers will compare PE male patients and healthy young men to see if PE posture defect affects postural stability.

DETAILED DESCRIPTION:
The experiment was designed as a pretest-posttest control trial. The clinical examination and surgery intervention (minimally invasive repair of pectus excavatum - MIRPE) of pectus excavatum patients are done in Wielkopolska Centre of Pulmonology and Thoracosurgery in Poznań, Poland. Other postural stability assessment of both, experimental group and control group subjects are done in the Poznań University of Physical Education in Poland. The measurements are carried out twice, before and three months after the intervention for experimental group, and twice for control group as well. Before the experiment initial measurements connected to basic and somatic characteristics assessments are recorded. Participants are also familiarized with measurement methods.

All PE patients included in the study after preoperative examination undergo the Nuss surgery procedure (MIRPE): curved metal bars are inserted behind the sternum to correct the shape of the anterior chest wall. The bars are left in situ for three years and then removed. The operation is performed under general anesthesia in a hospital setting.

Postural stability as a dependent variable was examined with the use of the posturography method based on the measurement of centre of pressure (COP) displacements. The stabilometric platform CQStab2P in two-plates version (CQ Electronic System, Poland) is used for collecting COP data during trials. The platforms are equipped with strain gauges that facilitated the monitoring of the changes in ground reaction forces. It is connected to a computer equipped with software provided by the manufacturer of the platforms. Based on the data of ground reaction forces the position and displacements of COP are estimated in the software.

The sampling frequency of 200 Hz is used during data acquisition. According to producer declaration processing accurancy is equal to 0.1% (12-bit processing, effective 10-bit) during reproduction of statokinesiogram with accurancy of 1 mm with radius fluctuation of 10cm.

The force platforms are placed on a hard and flat floor surface. Before the start of the testing procedures, the participants rest in a sitting position for 5 min. During the measurement, only the researcher and the participant are present in the room. Participants need to perform trials in three conditions: 1) double stance with eyes open (EO); 2) double stance with eyes closed (EC); 3) one-leg standing with eyes open (OLS).

Each trial is run two times - summing 6 trials in each measurement with a 20-second break between the following trials. The order of trials is random to avoid potential learning effects. An average of two repetitions of specific trials is taken as the final result.

The primary outcomes of the study are:

1. Average velocity of COP displacements and its components in anterior-posterior (AP) and medio-lateral (ML) directions (Vavg, VavgAP, VavgML, respectively). It's calculated as a ratio of the total path length covered by COP during the trial, and the time of the trial (mm/s).
2. Indicators of the spatial distribution of COP displacements i.e.sway area (SA) and maximal COP displacementin AP and ML directions (MaxAP and MaxML, respectively). SA is calculated as the size of the area covered by the COP during the trial (mm2). MaxAP and MaxML are calculated as maximal swaydistance (mm) of the COP from the 0.0 point along Y and X axis in Cartesian coordinate system, respectively.

Study population is characterized also by age, body weight and height, and body mass index (BMI) - calculated as body weight/height2.

The main calculations related to the assessment of the variability of dependent variables are based on the ANOVA variance analysis method (test F). The analysis applied takes into account within-group factor of repeated measurements "time" with two levels (pre and post), and between-group factor "group" (experimental and control). For interaction effects ("group" × "time") the eta-squared effect size is calculated. The effect size indicates the percent of variance explained by particular effects of the dependent variable. To compare the average values of average velocities, area, and maximal COP displacement (both pre-post values within groups, and between groups in pre and post conditions) Bonferroni detailed post-hoc comparisons is used.

Between-groups comparison for secondary outcomes in pretest is done with the use of t-Student test. The minimum level of statistical significance was defined as p ≤ 0.05. The study is conducted using the Statistica v. 13.0 software program.

ELIGIBILITY:
Inclusion Criteria:

* pectus excavatum (experimental group)
* no posture defects (control group)
* no neurological disorders
* consent to the surgical intervention procedure (experimental group)

Exclusion Criteria:

* co-existence of defects in the anterior chest wall other than pectus excavatum
* presence of musculoskeletal anomalies

Min Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Postural Stability | Three months
  Postural stability as a dependent variable examined with the use of the posturography method based on the measurement of Centre of Pressure displacements.

SECONDARY OUTCOMES:
BMI | Single measurement
  Body mass index (BMI) - calculated as body weight/height2

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Jarosz, M.Sc., Principal Investigator — Poznan University of Physical Education
Locations (2):
- Poland (2):
  - Wielkopolska Centre of Pulmonology and Thoracic Surgery in Poznan, Poznan
  - Poznan University of Physical Education, Poznan

IPD SHARING:
Plan to Share IPD: Yes
Data files will be made available as supplementary files in the scientific publication. Personal data will not be disclosed, only the raw results of posturographic analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available as soon as the scientific article will be published.
Access Criteria: Access criteria will depend on the publisher of the scientific article.

REFERENCES:
- [Background] Pawlak K, Gasiorowski L, Gabryel P, Galecki B, Zielinski P, Dyszkiewicz W. Early and Late Results of the Nuss Procedure in Surgical Treatment of Pectus Excavatum in Different Age Groups. Ann Thorac Surg. 2016 Nov;102(5):1711-1716. doi: 10.1016/j.athoracsur.2016.04.098. Epub 2016 Jun 30. PMID 27373189
- [Background] de Loos ER, Daemen JHT, Pennings AJ, Heuts S, Maessen JG, Hulsewe KWE, Vissers YLJ. Minimally invasive repair of pectus excavatum by the Nuss procedure: The learning curve. J Thorac Cardiovasc Surg. 2022 Mar;163(3):828-837.e4. doi: 10.1016/j.jtcvs.2020.11.154. Epub 2020 Dec 10. PMID 33478832
- [Background] Blaszczyk JW, Beck M, Sadowska D. Assessment of postural stability in young healthy subjects based on directional features of posturographic data: vision and gender effects. Acta Neurobiol Exp (Wars). 2014;74(4):433-42. doi: 10.55782/ane-2014-2006. PMID 25576974